CLINICAL TRIAL: NCT05718934
Title: A Randomized Clinical Study to Compare Low Dose of Sugammadex to Standard Dose of Neostigmine and Glycopyrrolate for the Reversal of Rocuronium Induced Moderate Neuromuscular Block
Brief Title: Low Dose of Sugammadex vs Neostigmine and Glycopyrrolate for the Reversal of Rocuronium
Acronym: SUGANEO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Philippe Richebe, Director of Research, Principal Investigator, Anesthesiologist, Associate Professor, MD, PhD, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-3091
Record Dates: First submitted 2022-11-01; First posted 2023-02-08 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Neuromuscular Blockade
Keywords: sugammadex; neostigmine; general anesthesia
MeSH Terms: interventions — Neostigmine; Glycopyrrolate; Sugammadex

STUDY DESIGN:
Intervention Model Description: Two groups of patients randomized into Group "N" for neostigmine and group "S" for sugammadex for a total of 144 participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Two groups of patients randomized into Group "N" for neostigmine and group "S" for sugammadex. Group N will receive the standard reversal (neostigmine 50 µg.kg-1 and glycopyrrolate 7 µg.kg-1) and group S will receive sugammadex 0.5 mg.kg-1. Randomization will be done prior to the entrance in the OR, the day of the surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group "N" for Standard reversal (Active Comparator): Standard reversal of 50 µg.kg-1 neostigmine (up to a maximum dose of 5mg) and 7 µg.kg-1 glycopyrrolate at the end of surgery (when surgeons finish deep tissues closure) with starting TOF 1-3.
  Interventions: Drug: Neostigmine and glycopyrrolate
- Group "S" for Sugammadex (Experimental): Sugammadex 0.5 mg.kg-1 IV will be performed at the end of surgery (when surgeons finish deep tissues closure) with starting TOF 1-3.
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Neostigmine and glycopyrrolate — See arm descriptions
  Arms: Group "N" for Standard reversal
Drug: Sugammadex — See arm descriptions
  Arms: Group "S" for Sugammadex

SUMMARY:
The aim of this study is to compare the use of a low dose sugammadex and neostigmine combined to glycopyrrolate to reverse a rocuronium induced moderate neuromuscular blockade.

DETAILED DESCRIPTION:
Neuromuscular blocking agents (NMBAs) are administered by anesthesiologists for general anesthesia to facilitate endotracheal intubation and/or surgical conditions. Unfortunately, postoperative residual neuromuscular blockade (rNMB), is an adverse event usually observed after extubation in the postanesthesia care unit (PACU) after surgery. rNMB is associated with upper airway obstruction, reduced pharyngeal muscle coordination, decreased functional residual capacity, and impaired hypoxic ventilatory response and may lead to critical cardiopulmonary complications.To prevent those complications, monitoring NMBAs activity as well as appropriate reversal are crucial.

In the light of the strong evidence proving the superiority of sugammadex for the reversal of NMB, the investigators chose to examine whether a quarter dose (0.5 mg.kg-1) of sugammadex would be superior to neostigmine for the reversal of moderate NMB (TOF 1 to 3). The investigators believe that this strategy will encourage the routine use of sugammadex because of a drastically reduced cost per patient with an increased safety and less adverse events compared to neostigmine reversal.

This study will be conducted in a single center, double blinded, randomized controlled study.

Type of surgery: any surgery under general anesthesia in ASA 1-3 patients, fully consented.

In the OR, the investigators will place a standardized monitoring: ECG, non-invasive blood pressure and SpO2. The investigators will monitor the depth of anesthesia using the BIS index (Medtronic, Canada) and the intraoperative nociception balance using the NOL index (Medasense Ltd., Ramat Gan, Israel). Finally, the investigators will monitor neuromuscular blockade using TOF-scan® (Draeger, Mississauga, Canada). The stimulation electrodes will be placed on the forearm of the patient to monitor the response to ulnar stimulation of the adductor pollicis muscle.

The investigators will use adjusted body weight for the administration of the drugs used in our anesthesia protocol except for rocuronium, sugammadex and neostigmine that will be given based on the real actual body weight.

The primary objective of the study:

To compare the mean time for recovery of the TOF ratio to 0.9 (90%) at the end of the surgery for rocuronium induced moderate neuromuscular blockade (TOF 1 to 3 at the end of the surgery) in two groups: Group "N" for neostigmine and group "S" for sugammadex. Group N will receive the standard reversal (neostigmine 50 µg.kg-1 and glycopyrrolate 7 µg.kg-1) and group S will receive sugammadex 0.5 mg.kg-1.

Secondary objectives are listed below.

Based on a 2-sided alpha < 0.05 and 80% power, the investigators calculated that 64 patients per group was required to detect a clinically relevant effect size of 0.5 favouring S group. The sample size will be inflated to 144 (72 per group) to account for 10% withdrawals and loss of follow-up.

Study Duration: 12 months.

Study Center: Maisonneuve-Rosemont Hospital, CIUSSS de l'Est de l'Ile de Montreal (CEMTL), University of Montreal, Montreal, Quebec, Canada.

Adverse Events: None expected.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3 patients,
* Undergoing general anesthesia with rocuronium induced NMB,
* TOF 1-3 at the end of surgery,
* BMI < 36 kg.m-2,
* Age > 18 years old

Exclusion Criteria:

* History of coronary artery disease and unstable before surgery
* History of serious cardiac arrhythmia (including atrial fibrillation)
* Renal or hepatic dysfunction
* Obstructive sleep apnea requiring continuous positive airway pressure (CPAP) machine
* Neuromuscular disease
* Allergy to any drug used in the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Time for recovery from moderate NMB | Intra-operative (from T0 = incision until Tend = start dressing)
  Time, in minutes, for recovery of the TOF ratio to 0.9 at the end of the surgery for rocuronium induced moderate neuromuscular blockade (TOF 1 to 3 at the end of the surgery).

SECONDARY OUTCOMES:
Time for awakening and extubation | Intra-operative (from T0 = incision until Tend = start dressing)
  The time, in minutes for awakening and extubation. Time for awakening will start at the injection of the reversal agent and end when the patient is opening his eyes. Time for extubation will start at the same time point and will end when extubation is complete.
Incidence of reoccurrence of NMB | Intra-operative (from T0 = incision until Tend = start dressing)
  The incidence of rNMB (defined as TOF ratio < 0.9 30 min after the end of reversal agent administration) and the incidence of NMB reoccurrence (defined as a decrease in TOF ratio from ≥ 0.9 to < 0.8 for at least 3 consecutive TOF values)
Incidence of critical respiratory event | Every 15 minutes until discharge from PACU, up to 2 hours
  The incidence of critical respiratory event (CRE). A CRE will be defined as the occurrence of one of the following criteria:
  * Upper airway obstruction requiring an intervention
  * Moderate hypoxemia: SpO2 of 90-93% on 2 L.min-1 nasal cannula O2 that was not improved after active interventions
  * Severe hypoxemia: SpO2 < 90% on 2 L.min-1 nasal cannula O2 that was not improved after active interventions
  * Signs of respiratory distress or impeding ventilatory failure
  * Inability to beath deeply when requested to by a PACU nurse
  * Patient complaining of symptoms of respiratory or upper airway muscle weakness
  * Patient requiring reintubation in the PACU
  * Clinical evidence or suspicion of pulmonary aspiration after tracheal extubation
Vital signs changes - Mean arterial pressure | Every 15 minutes until discharge from PACU, up to 2 hours
  Difference between pre-reversal values and values for mean arterial pressure (mmHg) obtained 2, 5, 10 and 30 min after reversal.
Vital signs changes - Heart rate | Every 15 minutes until discharge from PACU, up to 2 hours
  Difference between pre-reversal values and values for heart rate (bpm) obtained 2, 5, 10 and 30 min after reversal.
Vital signs changes - Oxygen saturation | Every 15 minutes until discharge from PACU, up to 2 hours
  Difference between pre-reversal values and values for SpO2 (%) obtained 2, 5, 10 and 30 min after reversal.
Vital signs changes - Respiratory rate | Every 15 minutes until discharge from PACU, up to 2 hours
  Difference between pre-reversal values and values for respiratory rate (respiration per minute) obtained 2, 5, 10 and 30 min after reversal.
PACU scores - Aldrete | Every 15 minutes until discharge from PACU, up to 2 hours
  Difference in Aldrete's score at rest between group and time to reach scores to discharge between groups.
  5 criterias : I-Consciousness level II-Respiration III- Hemodynamics IV-Motricity V- Oxygen saturation
  Minimum score : 0 Maximum score : 10
PACU scores - Maisonneuve-Rosemont PACU score | Every 15 minutes until discharge from PACU, up to 2 hours
  Difference in Maisonneuve-Rosemont PACU score at rest between groups and time to reach scores to discharge between groups.
  8 criterias : I-Consciousness level II-Respiration III- Hemodynamics IV-Motricity V- Oxygen saturation VI- Pain VII- Nausea/Vomiting VIII- Surgical bleeding
  Minimum score : 0 Maximum score : 16
PACU scores - PONV score | Every 15 minutes until discharge from PACU, up to 2 hours
  Difference in Postoperative nausea and vomiting (PONV) score at rest between groups and time to reach scores to discharge between groups.
  0- No nausea/vomiting
  1. Nausea without the need of a treatment
  2. Nausea needing a treatment
  3. Nausea and vomiting
PACU scores - POSS score | Every 15 minutes until discharge from PACU, up to 2 hours
  Difference in Pasero Opioid-induced Sedation Scale (POSS) score at rest between groups and time to reach scores to discharge between groups.
  S- Normal sleep easy awakening
  1. Awake and alert
  2. Sometimes drowsy, easy awakening
  3. Drowsy, wakes up but falls asleep during conversation
  4. Sleeps soundly, wakes up with difficulty or not at all to stimulation
PACU scores - NRS pain score | Every 15 minutes until discharge from PACU, up to 2 hours
  Difference in Nnumeric Rating Scale (NRS) pain score at rest between groups and time to reach scores to discharge between groups.
  Scale between 0 meaning "no pain" and 10 meaning "the worst pain imaginable"
Time spent in PACU | Every 15 minutes until discharge from PACU, up to 2 hours
  Total time, in minutes spent in PACU
Cost of reversal agent | Intra-operative (from T0 = incision until Tend = start dressing)
  Cost, in CAD, associated with reversal agent
Overall cost | Intra-operative (from T0 = incision until Tend = start dressing) to PACU discharge, up to 2 hours
  Cost evaluation, in CAD, associated with extubation time in the operating room and PACU stay.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe PR Richebé, MD PhD, Principal Investigator — CIUSSS Est de l'île de Montréal
Locations (1):
- CIUSSS de l'Est de l'Ile de Montreal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Hadj-Mimoune S, Morisson L, Ellassraoui S, Idrissi M, Quach M, Godin N, Oulehri W, Fortier LP, Verdonck O, Laferriere-Langlois P, Richebe P. Low dose of sugammadex versus neostigmine for reversal of rocuronium induced moderate neuromuscular block: a randomized controlled trial. BMC Anesthesiol. 2026 Jan 17. doi: 10.1186/s12871-025-03581-2. Online ahead of print. PMID 41545820